CLINICAL TRIAL: NCT05125471
Title: COBI-AVM Study - Phase 2 Study to Assess the Safety and Efficacy of Cobimetinib In Extracranial Arteriovenous Malformations (AVM)
Brief Title: Cobimetinib In Extracranial Arteriovenous Malformations (COBI-AVM Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 261983
Record Dates: First submitted 2021-11-12; First posted 2021-11-18 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-06

CONDITIONS: Arteriovenous Malformations (Extracranial)
MeSH Terms: conditions — Arteriovenous Malformations | interventions — cobimetinib

STUDY DESIGN:
Intervention Model Description: Cobimetinib will be given orally at the recommended phase 2 dose (RP2D).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Investigational Drug (Experimental): Cobimetinib will be administered at a maximal dose of 60 mg daily for 21 days on, then 7 days off, in a 28-Day treatment cycle for 12 cycles (approximately 12 months). Cobimetinib should be taken once daily at approximately the same time each day, and no later than 4 hours after the scheduled time. Cobimetinib can be taken with or without a meal. Cobimetinib tablets should never be chewed, cut, or crushed. Therapy may continue for up to 12 cycles provided the subject meets the criteria for starting subsequent cycles and does not meet any of the criteria for cobimetinib discontinuation. At least 7 days off cobimetinib (within +7 days) is required prior to starting a new treatment cycle.
  Interventions: Drug: Cobimetinib

INTERVENTIONS:
Drug: Cobimetinib — Adult dosing (>/= 18 years old) will be 60 mg orally once daily (tablet formulation); Pediatric dosing (<18 years old) will be 1 mg/kg/dose (maximum 60 mg per dose) orally once daily (oral suspension formulation).
  Other Names: Cotellic

SUMMARY:
The purpose of this open-label study is to evaluate the safety and efficacy of cobimetinib in extracranial AVM.

DETAILED DESCRIPTION:
After being informed of the study and potential risks, all patients giving informed consent will go undergo a screening period to determine eligibility for study entry. Patients who meet the eligibility requirements will be given cobimetinib to take by mouth once daily at the same time each day for 21 days and then have 7 days with no treatment. Patients will receive cobimetinib as a tablet (adult) or as a liquid (child).

ELIGIBILITY:
Inclusion Criteria:

* 2 years to 80 years of age
* Extracranial AVM with volumetric measurable disease AVM Tissue from a prior biopsy along with the corresponding pathology report will be required. If not available, a biopsy will be performed per standard of care
* Patient must be able to take an enteral dose and formulation of medication. Study medication is only available as an oral suspension or tablet, which may be taken by mouth or other enteral route such as nasogastric or gastric tube
* Karnofsky ≥ 50% for patients > 16 years of age and Lansky ≥ 50% for patients ≤ 16 years of age
* ANC ≥ 0.75 x 109/L (unsupported/without growth factor stimulant in past 7 days) Platelet count ≥ 75 x 109/L (unsupported/without transfusion in past 7 days) Hemoglobin ≥ 8 g/dL (unsupported/without transfusion in past 7 days)
* Calculated creatinine clearance (or radioisotope GFR) ≥ 70 mL/min/1.73m2 or serum creatinine based on age/gender as follows:

  * Age 2 < 6 years: Male 0.8; Female 0.8
  * Age 6 to < 10 years: Male1; Female 1
  * Age 10 to < 13 years: Male 1.2; Female 1.2
  * Age 13 to < 16 years: Male 1.5; Female 1.4
  * Age >/= 16 years: Male 1.7; Female 1.4
* AST and ALT ≤ 2.5 x upper limit of normal (ULN) for age Bilirubin (sum of conjugated + unconjugated) ≤ 1.5 x ULN for age
* Fractional shortening (FS) of ≥ 30% or ejection fraction of ≥ 50% by echocardiogram (ECHO) at Baseline, as determined by echocardiography within 21 days prior to study entry
* Female patients of childbearing potential (FOCBP) require a negative urine or serum pregnancy test at Baseline, within one week prior to the start of each cycle, at the End of Treatment (EOT) visit, and at the 28-Day Post-Treatment Safety Follow-Up (Safety Follow-Up) visit
* Female patients of childbearing potential and female partners of male patients who are pregnant or could become pregnant (i.e., females childbearing potential) must agree to follow the contraceptive requirements using two forms of effective contraceptive methods (one of which must be a barrier method) for the duration of the study treatment and for at least 3 months after the last dose of cobimetinib to avoid pregnancy and/or potential adverse effects on a developing embryo. Agreement to true abstinence (not periodic abstinence or withdrawal method) is an acceptable method of birth control
* Patients must also agree not to donate eggs (female patients) or sperm (male patients) during this study and for at least 3 months after the last dose of cobimetinib

Exclusion Criteria:

* Patients taking strong inducers or inhibitors of CYP3A4 within 14 days prior to study entry, including but not limited to erythromycin, clarithromycin, ketoconazole, azithromycin, itraconazole, grapefruit juice, or St. John's Wort. Appendix A includes a list of other known CYP3A4 inducers and inhibitors that should be discontinued at least 14 days prior to initiation of cobimetinib and avoided during study participation, if reasonable alternatives exist
* Completion of previous chemotherapy, immunotherapy, or targeted therapy for extracranial AVM with resolution of all associated toxicity to ≤ Grade 1 (except for alopecia and ototoxicity, which do not need to be resolved ≤ Grade 1) at least 28 days prior to study entry (except if otherwise specified below). Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to study entry. If, after the required timeframe, the laboratory eligibility criteria are met, the patient is considered to have recovered adequately
* Treatment with a long-acting hematopoietic growth factor within 14 days prior to initiation of cobimetinib or a short-acting hematopoietic growth factor within 7 days prior to study entry
* Treatment with hormonal therapy (except hormone replacement therapy or oral contraceptives), immunotherapy, biologic therapy, investigational therapy, or herbal cancer therapy within 28 days or < 5 half-lives, whichever is longer, prior to study entry
* Corticosteroid therapy < 0.5 mg/kg/day averaged during the month prior to study entry is permissible but must be discontinued 14 days prior to study entry
* Active malignancy or history of secondary malignancy
* History of severe hypersensitivity reactions to components of cobimetinib
* Refractory nausea and vomiting, malabsorption, external biliary shunt
* Patients who have a known active infection (excluding documented fungal infection of the nail beds) within 28 days prior to study entry that has not completely resolved
* Major surgical procedure or significant traumatic injury within 28 days prior to study entry, or anticipation of the need for major surgical procedure during the course of the study. Placement of a vascular access device or minor surgery is permitted within 14 days of study entry (provided the wound has healed)
* History of significant bowel resection that would preclude adequate absorption or other significant malabsorptive disease
* History of pneumonitis
* Ophthalmologic considerations: Patients with known significant ophthalmologic conditions or known risk factors for retinal vein occlusion are not eligible. Specifically, patients with a history of retinal vein occlusion (RVO), retinal detachment, retinal pathology on ophthalmologic exam, retinopathy of prematurity, central serous chorioretinopathy (CSSCR), neovascular retinopathy, intraocular pressure > 21 mmHg, and predisposing factors to RVO (e.g., uncontrolled hypertension, diabetes, or hyperlipidemia, coagulopathy) will be excluded
* Any other disease, metabolic or psychological dysfunction, physical examination or clinical laboratory finding giving reasonable suspicion of a disease or condition that in the opinion of the Investigator's judgement contraindicates use of an investigational drug or places the patient at unacceptable risk from treatment complications
* Clinically significant cardiac arrhythmias or unstable arrhythmia including bradyarryhthmias and/or patients who require anti-arrhythmic therapy (with the exception of beta-blockers or digoxin). Patients with controlled atrial fibrillation are not excluded.
* Unstable angina, or new-onset angina within 3 months prior to initiation of cobimetinib
* Symptomatic congestive heart failure, defined as New York Heart Association Class II or higher
* Myocardial infarction within 3 months prior to initiation of cobimetinib
* Known chronic human immunodeficiency virus (HIV)
* History of ≥ Grade 2 central nervous system (CNS) hemorrhage or history of any CNS hemorrhage within 28 days of study entry
* Female patients who are pregnant or lactating. Pregnant or lactating women will not be enrolled in this study because there is no available information regarding human fetal or teratogenic toxicities.
* Patient has received treatment with investigational therapy within 4 weeks prior to initiation of cobimetinib.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
Complete response (CR) or partial response (PR) rate compared to Baseline | Through study completion, an average of 1 year
  Response will be determined by a blinded, centralized review of volumetric MRI. Partial response is defined as a >/= 20% reduction in target extracranial AVM volume

CONTACTS AND LOCATIONS:
Overall Officials: Joana M Mack, MD, Principal Investigator — University of Arkansas for Medical Sciences, Arkansas Children's Hospital; Kevin J Bielamowicz, MD,, Principal Investigator — University of Arkansas for Medical Sciences, Arkansas Children's Hospital
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No